CLINICAL TRIAL: NCT03986320
Title: A Multi-site, Interventional, Comparative, Single-arm Trial to Evaluate the Safety and Effectiveness of Keeogo™ Dermoskeleton in Subjects With Hemiparesis Due to Ischemic or Hemorrhagic Stroke.
Brief Title: Evaluation of the Effectiveness and Safety of Keeogo™ Dermoskeleton in Subjects With Mobility Impairments Due to Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: B-Temia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KEOG-SE-002
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Stroke; Hemiparesis; Cerebral Vascular Accident
Keywords: Keeogo™; Dermoskeleton; Powered dermoskeleton; Lower limb dermoskeleton; Assistive exoskeleton; Orthotic dermoskeleton
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Device: Keeogo™ Dermoskeleton This device is intended for use in rehabilitation institutions to assist individuals with hemiparesis due to stroke who are able to stand and initiate a step in performing ambulatory functions.
Masking Description: Sites will enroll participants in order of recruitment. No other randomization procedure will be applied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Keeogo™ Dermoskeleton (Experimental): Keeogo™ Dermoskeleton is a low-profile, assistive exoskeleton (or 'dermoskeleton') that orthotically fits to the lower limbs. Keeogo™ is worn on the user's lower body using a belt and contact areas attached around the thighs and calves.
  Interventions: Device: Keeogo™ Dermoskeleton

INTERVENTIONS:
Device: Keeogo™ Dermoskeleton — This device is intended for use in rehabilitation institutions to assist individuals with hemiparesis due to stroke who are able to stand and initiate a step in performing ambulatory functions.

SUMMARY:
A multi-site, interventional, non-comparative, single-arm trial to evaluate the safety of the Keeogo™ Dermoskeleton in subjects with hemiparesis due to ischemic or hemorrhagic stroke.

DETAILED DESCRIPTION:
Stroke affects thousands of individuals annually, leading to considerable physical impairment and functional disability. Gait is one of the most important activities of daily living affected in this patient population. Recent technological developments in passively powered dermoskeleton can create powerful adjunctive tools for rehabilitation and potentially accelerate functional recovery. Here, the investigators present the development and evaluation of a lower limb dermoskeleton, namely Keeogo™ (B-Temia), for use in rehabilitation institutions to assist individuals with hemiparesis due to stroke who are able to stand and initiate a step in performing ambulatory functions.

Keeogo™ Dermoskeleton is a low-profile, assistive exoskeleton (or 'dermoskeleton') that orthotically fits to the lower limbs. Keeogo™ is worn on the user's lower body using a belt and contact areas attached around the thighs and calves.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Provide signed and dated informed consent form;
* Willing to comply with all study procedures and be available for the duration of the study [2-3 days per week, 3-5 consecutive weeks];
* Adults 18 years of age and older;
* Confirmed Cerebrovascular Accident (CVA) with hemiparesis;
* Stable stroke (≥ 6 months post-incident)
* Sufficient cognition to follow simple instructions and understand the content and purpose of the study (MMSE > 20);
* Capable of standing and walking independently for an extended period of time (MMT

  * 3 hip flexors and extensors, and ≥ 2 knee flexors and extensors with BBS ≥ 45);
* Presence of any gait deficit, as defined by one or more of the following clinical observations:

  * Hip hike
  * Hip circumduction
  * Knee spasticity (MAS 2 to 3) as per Modified Ashworth Scale (MAS)
  * Mid-foot striking (aka 'flat foot landing')
  * Poor foot clearance (toe/foot drop or foot drag)
  * Narrow steps (< 1 shoe-width or < 8 cm)
* Manual Muscle Test (MMT) of 4/5 for the unaffected upper extremity;
* Able to sit on a bench for more than 5 minutes;
* Is physically and mentally compatible with device to demonstrate ability to safely activate the Keeogo™ user interface;
* Able to understand and follow instructions with assistance if needed.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Legally blind
* Pregnant, lactating, or postpartum sacroiliac joint recovery is ongoing (recent childbirth, not yet cleared for vigorous exercise)
* Skin condition that contraindicates use of orthotics or support braces
* Recent (<6 mo) lower-body hospitalizations or active treatments due to a joint, muscle, bone, nerve or vascular injury or condition
* Scheduled for major surgery within next 4 months
* Lower-extremity amputation above or below the knee
* Have uncontrolled hypertension
* Recent (<1 year) heart attack
* Have uncontrolled diabetes
* Diagnosed with other health condition(s) that affect mobility and balance; chronic obstructive pulmonary disease; peripheral arterial disease; vestibular disorders; cerebellar disease; cerebral palsy; muscular dystrophy spinal cord injury; other brain injury aside from the reported CVA;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related adverse events [Safety] | Duration of study participation for each subject, estimated 3-5 weeks
  Safety will be evaluated on the basis of the number of device-related serious adverse events reported for subjects during their participation in the study.

SECONDARY OUTCOMES:
Incidence of device malfunctions during study procedures [Device Reliability] | Duration of study completion for each site, estimated 3-5 weeks
  Device reliability will be evaluated on the basis of the number of device malfunctions reported by research study staff for the duration of study procedures at each study site.
Incidence of injury to Physical Therapist (PT) caused by device [PT safety] | Duration of study completion for each site, estimated 3-5 weeks
  PT safety will be evaluated on the basis of the number of serious device-related injuries reported by study physical therapists for the duration of study procedures at each study site.
Device, Effectiveness | Duration of study participation for each subject, estimated 3-5 weeks
  Clinician and Patient Reported Outcomes (surveys) will be used to assess the effectiveness of the device in assisting gait. The surveys will rate subject performance in walking based on clinician observed deviations and subject perception of mobility limitation due to the stroke.
  * Device effectiveness will be measured based on statistical analysis of the survey data between conditions (baseline compared to device-use) Ratings by the surveys will be validated using instrumented walkway and image data collected during walking.

OTHER OUTCOMES:
30-Second Chair Stand Test | Duration of study completion for each site, estimated 3-5 weeks
  Subjects sit in the middle of chair and place hands on opposite shoulder crossed at wrists. Keeping feet flat on floor, back straight, arms against chest, subjects rise to full standing position when told "go" followed by sit down, the start position. This movement is repeated for as many times as possible for 30 seconds. Additionally, the test is repeated for a total of 5 cycles with short rest (≤ 90 seconds) between sets.
  Patient and Clinician reported outcomes are assessed for this measure via a sit-to-stand-to-sit question on the survey given for the secondary effectiveness endpoint.
Timed Stair Test | Duration of study completion for each site, estimated 3-5 weeks
  Subjects start with both feet on the bottom landing then ascend and descend a set number of stairs as quickly as possible in a safe manner using a rail only if needed. Time is recorded from ascent through descent.
  Patient and Clinician reported outcomes are assessed for this measure via a stair ascent/descent question on the survey given for the secondary effectiveness endpoint.
Patient and Clinician Reported Outcomes (surveys) | Duration of study completion for each site, estimated 3-5 weeks
  Questionnaires provide patient and clinician-centric view of treatment of gait deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD., Principal Investigator — Shirley Ryan Ability Lab (SRA)
Locations (4):
- United States (3):
  - Shirley Ryan Ability Lab (SRA), Chicago, Illinois
  - Human Performance and Engineering Research (HPER), West Orange, New Jersey
  - James J Peters VA Medical Center - Center for the Medical Consequences of Spinal Cord Injury, The Bronx, New York
- Assistive Technology Clinic (ATC), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buesing C, Fisch G, O'Donnell M, Shahidi I, Thomas L, Mummidisetty CK, Williams KJ, Takahashi H, Rymer WZ, Jayaraman A. Effects of a wearable exoskeleton stride management assist system (SMA(R)) on spatiotemporal gait characteristics in individuals after stroke: a randomized controlled trial. J Neuroeng Rehabil. 2015 Aug 20;12:69. doi: 10.1186/s12984-015-0062-0. PMID 26289955
- [Background] Xu J, Murphy SL, Kochanek KD, Bastian B, Arias E. Deaths: Final Data for 2016. Natl Vital Stat Rep. 2018 Jul;67(5):1-76. PMID 30248015
- [Background] He Y, Eguren D, Luu TP, Contreras-Vidal JL. Risk management and regulations for lower limb medical exoskeletons: a review. Med Devices (Auckl). 2017 May 9;10:89-107. doi: 10.2147/MDER.S107134. eCollection 2017. PMID 28533700
- [Background] Lee SH, Lee HJ, Chang WH, Choi BO, Lee J, Kim J, Ryu GH, Kim YH. Gait performance and foot pressure distribution during wearable robot-assisted gait in elderly adults. J Neuroeng Rehabil. 2017 Nov 28;14(1):123. doi: 10.1186/s12984-017-0333-z. PMID 29183379
- [Background] Morawietz C, Moffat F. Effects of locomotor training after incomplete spinal cord injury: a systematic review. Arch Phys Med Rehabil. 2013 Nov;94(11):2297-308. doi: 10.1016/j.apmr.2013.06.023. Epub 2013 Jul 9. PMID 23850614
- See also: Disability and Functioning (Noninstitutionalized Adults Aged 18 and Over) — https://www.cdc.gov/nchs/fastats/disability.htm
- See also: Mapping Connections. An Understanding of Neurological Conditions in Canada. The National Population Health Study of Neurological Conditions.: Neurological Health Charities Canada. Government of Canada. Canadian Institutes of Health Research. — http://www.phac-aspc.gc.ca/publicat/cd-mc/mc-ec/assets/pdf/mc-ec-eng.pdf
- See also: Canada S. Canada at a Glance 2018. Population — https://www150.statcan.gc.ca/n1/pub/12-581-x/2018000/pop-eng.htm
- See also: Medical Devices; Physical Medicine Devices; Classification of the Powered Exoskeleton A Rule by the Food and Drug Administration on 02/24/2015 — https://www.federalregister.gov/documents/2015/02/24/2015-03692/medical-devices-physical-medicine-devices-classification-of-the-powered-exoskeleton
- See also: (CDC) CfDCaP. National Center for Health Statistics - Cerebrovascular Disease or Stroke — https://www.cdc.gov/nchs/fastats/stroke.htm